CLINICAL TRIAL: NCT03965325
Title: FOcUs on Colorectal CAncer oUtcomes: Long-Term Study
Acronym: Foucault
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Other Study IDs: 19-001
Record Dates: First submitted 2019-05-03; First posted 2019-05-29 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
Keywords: Value-Based Health Care; VBHC; Patient reported outcomes measure; PROMs; PROs; Colorectal Cancer; Patient reported outcomes
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Use of a standardized set to collect clinical and patient-centered data, to assess the trend of the Global Health Status overtime in colorectal cancer patients — Patients' data (baseline characteristics, clinical and PROMs outcomes) will be collected according to patient-centered standardized set regarding ICHOM recommendations. Data collection and the follow-up schedule are carried out at : baseline (before any treatment or surgery), 1- and 6-month follow-up and then once a year.

SUMMARY:
Colorectal cancer (CRC) affects men and women of all racial and ethnic groups and accounts for more than 600,000 deaths per year, globally. Current treatment options may involve surgery, chemotherapy (both adjuvant and neoadjuvant), radiation therapy, and palliative care, each with trade-offs between disease management and patients' quality of life. Unfortunately, significant disparity exists in the quality of care and there is a need for standardization to ensure high-value health care for all patients.

This study evaluates the introduction of a Value-Based Health Care (VBHC) patient-centered framework in CRC treatments. VBHC is an innovative approach that aims to improve health care by identifying and systematically measuring both medical and patient-reported health care outcomes and costs. By applying sets of disease-specific outcomes measurements, health care providers (HCP) can compare care strategies and make informed choices with regard to optimization of care, necessary investments and possible cost reductions.

The adoption of a VBHC patient-centered approach may have a significant impact on therapeutic areas constituting a major disease and cost burden for the global health care, such as CRC. It has the potential to improve cancer care planning, monitoring, and management of patients, by promoting better communication and shared decision making by patients and HCP.

A patient-reported outcome measurement (PROM) is defined as any report about a health condition and its treatment that comes directly from the patient. The use of a tailored pathway including PROMs improve both quality of life (QoL) and survival in cancer patients. Another essential requirement of VBHC approach is the outcome monitoring, to allow HCP accessing to evidence-based, simplified information on the hospital clinical practice and potentially increase health value for both patients and HCP. For patients with CRC, the International Consortium for Health Outcomes Measurement (ICHOM) developed a comprehensive patient-centered outcomes measurement set that could be used in the clinical practice to monitor patients' status.

The purpose of this study is to evaluate the introduction of a VBHC approach in CRC treatments, using a validated VBHC set of clinical outcomes and PROMs, to understand which practice would be most effective in achieving patient-centered care. The underlying hypothesis is that a periodic analysis of these outcomes could increase health value for both patients and HCPs.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) affects men and women of all racial and ethnic groups and accounts for more than 600,000 deaths per year, globally. Current treatment options may involve surgery, chemotherapy (both adjuvant and neoadjuvant), radiation therapy, and palliative care, each with trade-offs between disease management and patients' quality of life. Unfortunately, significant disparity exists in the quality of care, and so outcomes delivered across institutions for each treatment modality, suggesting that unwarranted variation in the provision of care occurs for patients with CRC. Hence, there is a need for standardization to ensure high-value health care for all patients, regardless the hospital where they present.

This study evaluates the introduction of a Value-Based Health Care (VBHC) patient-centered framework in CRC treatments. VBHC is an innovative approach that aims to improve health care by identifying and systematically measuring both medical and patient-reported health care outcomes. By applying sets of disease-specific outcomes measurements, health care providers (HCP) can compare care strategies and make informed choices with regard to optimization of care, necessary investments and possible cost reductions. The need to move toward a more patient-centered approach has been highlighted to be crucial in the context of quality care. Patient-centered care is a key component of a health system that ensures that all patients have access to the outcomes that matter for them.

The adoption of a VBHC patient-centered approach may have a significant impact on therapeutic areas constituting a major disease and cost burden for the global health care, such as CRC. CRC causes significant morbidity and mortality, being the third most common cancer and the fourth most common cause of cancer deaths worldwide and the second most common cause of cancer deaths in Europe. The 5-years relative survival rate is 47% in Europe and 60% in the US. Moreover, the economic burden of CRC is expected to increase in the future, partly due to changing demographics and the introduction of new and resource-demanding treatments and screening methods. In this scenario, the introduction of VBHC-based clinical pathways has the potential to improve cancer care planning, monitoring, and management of patients, by promoting better communication and shared decision making by patients and healthcare providers.

Research Hypothesis In general, an essential requirement to be able to apply a VBHC approach is the clear definition of the disease-specific outcomes, both clinical and patient-reported. Clinical outcomes can be measured by activity data such as complication rates, type of surgery, re-hospitalization rates, or by agreed scales and other forms of measurement. A patient-reported outcome measurement (PROM) is defined as any report about a health condition and well-being (quality of life) that comes directly from the patient using a self-reported measure, without interpretation of the patient's response by a physician or anyone else.

PROMs are being advocated for use in routine clinical cancer practice and for the early detection of patient distress. The use of a tailored pathway including PROMs has been shown to improve both quality of life (QoL) and survival in cancer patients. The QoL, by assessing physical function and symptoms such as pain, and social functioning are known to be independent prognostic factors for overall survival of metastatic CRC patients.

Another essential requirement of VBHC approach is the outcome monitoring, to allow HCP accessing to evidence-based, simplified information on the hospital clinical practice and potentially increase health value for both patients and HCPs. It has been demonstrated that facilitation of data interpretation can improve medical care quality. In particular, a Dutch nationwide study showed that, by providing continuous feedback of benchmarked performance information to colorectal surgeons, clinical outcomes of patients undergoing colorectal cancer surgery improves and cost decreases.

For patients with CRC, the International Consortium for Health Outcomes Measurement (ICHOM) developed a comprehensive patient-centered outcomes measurement set that could be used in the clinical practice to monitor patients' status. Therefore, an exploratory study collecting ICHOM set of data could provide useful information to evaluate the feasibility, benefits and barriers of a VBHC approach for CRC.

The purpose of this study is then to evaluate the introduction of a VBHC approach in CRC treatments, using a validated VBHC set of clinical outcomes and PROMs, to understand which practice would be most effective in achieving patient-centered care. The underlying hypothesis is that a periodic analysis of these outcomes could increase health value for both patients and HCPs. The study will first explore the most accurate feasible trend of the Global Health Status (Quality of Life evolution) of patients but also clinical outcomes and other PROMs trends over time, the cause(s) of these trends, and whether any outcomes' predictors can be found. Furthermore, a general assessment of the impact of the VBHC approach on CRC treatments will be performed, in terms of general satisfaction and knowledge in medical care. Finally, cost associated with performed procedures and complications will be estimated ambispectively using the Time-driven Activity-based Costing (TDABC) methodology, where applicable. Additional participating sites shall be free to apply the same methodology or to measure costs derived from traditional hospital cost accounting systems.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed CRC diagnosis not older than 8 years from the first treatment;
2. Age ≥18 years or minimum age as required by local regulations;
3. Ability and willingness to give written consent form ("Patient informed consent Form" or "Patient Data Release Authorization Form");
4. Ability and willingness to comply with the clinical investigational plan.

Exclusion Criteria:

1. Pregnant or breastfeeding woman;
2. Psychiatric and cognitive impairment;
3. Patient under juristic protection or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with a CRC who had a surgical consultation, and who meet the inclusion/exclusion criteria are intended to participate in this study. Subject enrollment will continue for the whole study duration. The eligibility criteria are kept comprehensive to all CRC types to reflect centers routine clinical practice ("all-comer" or "real world" subjects). To avoid subject selection bias, consecutive screening and enrollment will be requested.
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Assess the most accurate trend of the Global Health Status (Quality of Life evolution) over time in colorectal cancer patients evaluated by the EORTC-QLQ-C30 questionnaire. | Baseline
  The EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire - C30) is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / Quality of Life (QoL) scale, and six single items.
  The global health status / Quality of Life scale runs from 1 (very poor) to 7 (excellent) and the others from 1 (not at all) to 4 (very much). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus:
  * a high score for a functional scale represents a high / healthy level of functioning,
  * a high score for the global health status / QoL represents a high QoL,
  * but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Assess the most accurate trend of the Global Health Status (Quality of Life evolution) over time in colorectal cancer patients evaluated by the EORTC-QLQ-C30 questionnaire. | Month 1 follow-up
  The EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire - C30) is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / Quality of Life (QoL) scale, and six single items.
  The global health status / Quality of Life scale runs from 1 (very poor) to 7 (excellent) and the others from 1 (not at all) to 4 (very much). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus:
  * a high score for a functional scale represents a high / healthy level of functioning,
  * a high score for the global health status / QoL represents a high QoL,
  * but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Assess the most accurate trend of the Global Health Status (Quality of Life evolution) over time in colorectal cancer patients evaluated by the EORTC-QLQ-C30 questionnaire. | Month 6 follow-up
  The EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire - C30) is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / Quality of Life (QoL) scale, and six single items.
  The global health status / Quality of Life scale runs from 1 (very poor) to 7 (excellent) and the others from 1 (not at all) to 4 (very much). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus:
  * a high score for a functional scale represents a high / healthy level of functioning,
  * a high score for the global health status / QoL represents a high QoL,
  * but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Assess the most accurate trend of the Global Health Status (Quality of Life evolution) over time in colorectal cancer patients evaluated by the EORTC-QLQ-C30 questionnaire. | Once a year, for maximum 3 years, from the second postoperative year
  The EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire - C30) is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / Quality of Life (QoL) scale, and six single items.
  The global health status / Quality of Life scale runs from 1 (very poor) to 7 (excellent) and the others from 1 (not at all) to 4 (very much). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus:
  * a high score for a functional scale represents a high / healthy level of functioning,
  * a high score for the global health status / QoL represents a high QoL,
  * but a high score for a symptom scale / item represents a high level of symptomatology / problems.

SECONDARY OUTCOMES:
Assess the trend of all VBHC outcomes (baseline characteristics, clinical and PROMs outcomes) over time in CRC patients by the EORTC-QLQ-C30 questionnaire | Baseline; Month 1 follow-up; Month 6 follow-up; Once a year, for maximum 3 years, from the second postoperative year
  The EORTC-QLQ-C30 questionnaire is composed of both multi-item scales and single-item measures:
  * the global health status score (Quality of Life), runs from 1 (very poor) to 7 (excellent);
  * the functional scores (Physical function, Emotional function, Anxiety…), runs from 1 (not at all) to 4 (very much).
  The trend of each category of PROMS given by the EORTC-QLQ-C30 will be evaluated in four groups of patients: tumor on the right and transverse part of the colon; tumor on the left part of the colon; rectal tumor; metastatic colorectal cancer.
Assess the trend of all VBHC outcomes (baseline characteristics, clinical and PROMs outcomes) over time in CRC patients by the EORTC-QLQ-CR29 questionnaire | Baseline; Month 1 follow-up; Month 6 follow-up; Once a year, for maximum 3 years, from the second postoperative year
  The symptom scores (Fatigue, Nausea and vomiting, Pain …), running from 1 (not at all) to 4 (very much), and given by EORTC (European Organisation for Research and Treatment of Cancer) will be evaluated by the use of the EORTC-QLQ-CR29 questionnaire.
  The trend of each category of PROMS given by the EORTC-QLQ-CR29 in four groups of patients: tumor on the right and transverse part of the colon; tumor on the left part of the colon; rectal tumor; metastatic colorectal cancer.
Assess the trend over time of the patient's baseline characteristics and outcomes regarding ICHOM (International Consortium for Health Outcomes Measurements) recommendations | Baseline; Month 1 follow-up; Month 6 follow-up; Once a year, for maximum 3 years, from the second postoperative year
  Trend over time will be analysed by means of Generalized Estimating Equation models as appropriate to account for repeated measures using patient as the subject. Baseline characteristics and outcomes will be assessed regarding ICHOM recommendations:
  * descriptive analysis of baseline characteristics (patients' demographic-, clinical-, tumor- and treatment factors, and treatment variables)
  * descriptive analysis of care status disutility (short-term treatment complications)
  * evaluation of the degree of health (Quality of Life, functioning, and long-term adverse effects) : from 1 (very poor) to 7 (excellent)
  * evaluation of the survival and disease control (number of overall survival, disease-specific survival, recurrence, and progression-free survival)
  * descriptive analysis of the quality of death (quality of end of life care (last 30 days of life))
  * evaluation of the symptoms score using EORTC-QLQ-C30 and CR29: from 1 (not at all) to 4 (very much)
Assess the proportion of missing clinical outcomes and PROMs data collected using the standardized set developed by the ICHOM for CRC | Baseline; Month 1 follow-up; Month 6 follow-up; Once a year, for maximum 3 years, from the second postoperative year
  The average number of missing clinical outcomes and PROMs data collected using the standardized set developed by the ICHOM for CRC at each follow-up visit will be calculated and used to determine the level of relevance and confidence for each variable
Assess the proportion of patients involved in this study compared to the whole cohort of patients who have been treated for a colorectal cancer at Strasbourg's University Hospital | Baseline; Month 1 follow-up; Month 6 follow-up; Once a year, for maximum 3 years, from the second postoperative year
  The proportion of patients involved in this study compared to the whole cohort of patients who have been treated for a colorectal cancer at Strasbourg's University Hospital and the proportion of patient who refused to participate to the study.
Assess the number of follow-up forms and their timelines | Baseline; Month 1 follow-up; Month 6 follow-up; Once a year, for maximum 3 years, from the second postoperative year
  The number of follow-up forms and their timelines, by patient
Assess the missing data pattern for each clinical outcomes and PROMs | Baseline; Month 1 follow-up; Month 6 follow-up; Once a year, for maximum 3 years, from the second postoperative year
  The outcomes and PROMs will be classified into the three main classes of missing pattern, i.e. univariate, monotone, and arbitrary, to select actions for future data collection
Investigate predictors of clinical and PROMs outcomes in a real-life context | Baseline; Month 1 follow-up; Month 6 follow-up; Once a year, for maximum 3 years, from the second postoperative year
  Predictors of clinical outcomes and PROMs will be investigated by performing univariate and multivariate statistical analysis, when appropriate
Assess the variation of clinical outcomes and PROMs | Baseline; Month 1 follow-up; Month 6 follow-up; Once a year, for maximum 3 years, from the second postoperative year
  Control charts will be used to monitor clinical outcomes and PROMs in both Variable data charts as individual, average and range charts and Combination Charts (x-bar standard deviation, process capability, etc.).
  Control charts will have the following features:
  * Data points could be averages of subgroup or individual measurements plotted on the x and y axis and joined by a line. Time is always on the x-axis.
  * The Average or Center Line is the average or mean of the data points and is drawn across the middle section of the graph.
  * The Upper Control Limit (UCL) is drawn above the centerline. This is equal to 3 or 2 times of the standard deviation line.
  * The Lower Control Limit (LCL) is drawn below the centerline. This is equal to 3 or 2 times of the standard deviation line.
Evaluate the impact of a VBHC approach on patients | Once a year, for maximum 3 years, from the second postoperative year
  The impact of a VBHC approach on patient will be qualitatively evaluated by collecting and analysing the annual survey responses from patients on their perception and satisfaction of a VBHC approach: scale from "very satisfied" to "not satisfied".
Evaluate qualitatively the impact of a VBHC approach on involved HCPs by collecting and analysing the annual interview responses from HCPs | Once a year, for maximum 3 years, from the second postoperative year
  The impact of a VBHC approach on HCPs will be qualitatively evaluated by collecting and analysing the annual interview responses from HCPs concerning the satisfaction (scale from "very satisfied" to "not satisfied"), the introduction of new recommendations during the follow-up period (e.g., addition or deletion of a specific follow-up visit) and knowledge in clinical practice (e.g., inclusion of pain specialists or psychologists). Survey data will be reported using summary statistics and supporting graphical representations.
Measure healthcare costs during the study period | Baseline; Month 1 follow-up; Month 6 follow-up; Once a year, for maximum 3 years, from the second postoperative year
  At the hepato-digestive pole, Strasbourg's University Hospital, healthcare costs will be measured by applying the Time-driven Activity-based Costing (TDABC) methodology. Other eventual additional participating sites will be free to apply the same methodology or to measure costs derived from traditional hospital cost accounting systems. An assessment of the outcomes of the two different approaches could be made between different methodologies

CONTACTS AND LOCATIONS:
Overall Officials: Didier Mutter, MD, PhD, Principal Investigator — Service Chirurgie Digestive et Endocrinienne, Nouvel Hôpital Civil de Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Zerillo JA, Schouwenburg MG, van Bommel ACM, Stowell C, Lippa J, Bauer D, Berger AM, Boland G, Borras JM, Buss MK, Cima R, Van Cutsem E, van Duyn EB, Finlayson SRG, Hung-Chun Cheng S, Langelotz C, Lloyd J, Lynch AC, Mamon HJ, McAllister PK, Minsky BD, Ngeow J, Abu Hassan MR, Ryan K, Shankaran V, Upton MP, Zalcberg J, van de Velde CJ, Tollenaar R; Colorectal Cancer Working Group of the International Consortium for Health Outcomes Measurement (ICHOM). An International Collaborative Standardizing a Comprehensive Patient-Centered Outcomes Measurement Set for Colorectal Cancer. JAMA Oncol. 2017 May 1;3(5):686-694. doi: 10.1001/jamaoncol.2017.0417. PMID 28384684
- [Background] van Zelm R, Coeckelberghs E, Sermeus W, De Buck van Overstraeten A, Weimann A, Seys D, Panella M, Vanhaecht K. Variation in care for surgical patients with colorectal cancer: protocol adherence in 12 European hospitals. Int J Colorectal Dis. 2017 Oct;32(10):1471-1478. doi: 10.1007/s00384-017-2863-z. Epub 2017 Jul 17. PMID 28717841
- [Background] Krell RW, Regenbogen SE, Wong SL. Variation in hospital treatment patterns for metastatic colorectal cancer. Cancer. 2015 Jun 1;121(11):1755-61. doi: 10.1002/cncr.29253. Epub 2015 Jan 29. PMID 25640016
- [Background] Kaplan RS, Porter ME. How to solve the cost crisis in health care. Harv Bus Rev. 2011 Sep;89(9):46-52, 54, 56-61 passim. PMID 21939127
- [Background] Efficace F, Innominato PF, Bjarnason G, Coens C, Humblet Y, Tumolo S, Genet D, Tampellini M, Bottomley A, Garufi C, Focan C, Giacchetti S, Levi F; Chronotherapy Group of the European Organisation for Research and Treatment of Cancer. Validation of patient's self-reported social functioning as an independent prognostic factor for survival in metastatic colorectal cancer patients: results of an international study by the Chronotherapy Group of the European Organisation for Research and Treatment of Cancer. J Clin Oncol. 2008 Apr 20;26(12):2020-6. doi: 10.1200/JCO.2007.12.3117. PMID 18421055
- [Background] Kriza C, Emmert M, Wahlster P, Niederlander C, Kolominsky-Rabas P. Cost of illness in colorectal cancer: an international review. Pharmacoeconomics. 2013 Jul;31(7):577-88. doi: 10.1007/s40273-013-0055-4. PMID 23636661
- [Background] Ekwueme DU, Howard DH, Gelb CA, Rim SH, Cooper CP. Analysis of the benefits and costs of a national campaign to promote colorectal cancer screening: CDC's screen for life-national colorectal cancer action campaign. Health Promot Pract. 2014 Sep;15(5):750-8. doi: 10.1177/1524839913519446. Epub 2014 Feb 6. PMID 24505055
- [Background] Van Cutsem E, Borras JM, Castells A, Ciardiello F, Ducreux M, Haq A, Schmoll HJ, Tabernero J. Improving outcomes in colorectal cancer: where do we go from here? Eur J Cancer. 2013 Jul;49(11):2476-85. doi: 10.1016/j.ejca.2013.03.026. Epub 2013 Apr 30. PMID 23642327
- [Background] Joranger P, Nesbakken A, Hoff G, Sorbye H, Oshaug A, Aas E. Modeling and validating the cost and clinical pathway of colorectal cancer. Med Decis Making. 2015 Feb;35(2):255-65. doi: 10.1177/0272989X14544749. Epub 2014 Jul 29. PMID 25073464
- [Background] Van Cutsem E, De Gramont A, Henning G, Rougier P, Bonnetain F, Seufferlein T. Improving Outcomes in Patients with CRC: The Role of Patient Reported Outcomes-An ESDO Report. Cancers (Basel). 2017 May 26;9(6):59. doi: 10.3390/cancers9060059. PMID 28587143
- [Background] Klinkhammer-Schalke M, Lindberg P, Koller M, Wyatt JC, Hofstadter F, Lorenz W, Steinger B. Direct improvement of quality of life in colorectal cancer patients using a tailored pathway with quality of life diagnosis and therapy (DIQOL): study protocol for a randomised controlled trial. Trials. 2015 Oct 14;16:460. doi: 10.1186/s13063-015-0972-y. PMID 26467994
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Keller DS, Stulberg JJ, Lawrence JK, Samia H, Delaney CP. Initiating statistical process control to improve quality outcomes in colorectal surgery. Surg Endosc. 2015 Dec;29(12):3559-64. doi: 10.1007/s00464-015-4108-y. Epub 2015 Feb 21. PMID 25701062
- [Background] McLean KA, Sheng Z, O'Neill S, Boyce K, Jones C, Wigmore SJ, Harrison EM. The Influence of Clinical and Patient-Reported Outcomes on Post-surgery Satisfaction in Cholecystectomy Patients. World J Surg. 2017 Jul;41(7):1752-1761. doi: 10.1007/s00268-017-3917-7. PMID 28280919
- [Background] Govaert JA, van Dijk WA, Fiocco M, Scheffer AC, Gietelink L, Wouters MW, Tollenaar RA. Nationwide Outcomes Measurement in Colorectal Cancer Surgery: Improving Quality and Reducing Costs. J Am Coll Surg. 2016 Jan;222(1):19-29.e2. doi: 10.1016/j.jamcollsurg.2015.09.020. Epub 2015 Nov 14. PMID 26721750
- [Background] Keel G, Savage C, Rafiq M, Mazzocato P. Time-driven activity-based costing in health care: A systematic review of the literature. Health Policy. 2017 Jul;121(7):755-763. doi: 10.1016/j.healthpol.2017.04.013. Epub 2017 May 10. PMID 28535996
- See also: ICHOM Colorectal cancer data collection reference guide — https://www.ichom.org/portfolio/colorectal-cancer/
- See also: Schön Klinik: Measuring Cost and Value — https://www.hbs.edu/faculty/Pages/item.aspx?num=41579
- See also: International Committee of Medical Journal Editors. Recommendations for the Conduct, Reporting, Editing, and Publication of Scholarly Work in Medical Journals — http://www.icmje.org/recommendations/